CLINICAL TRIAL: NCT04790305
Title: Effect of Huaier Granule on Postoperative Adjuvant Treatment for High-risk Early-stage Triple-negative Invasive Ductal Carcinoma: a Prospective, Multicenter, Randomized, Controlled, Open-label Study
Brief Title: Effect of Huaier Granule on Adjuvant Treatment for High-risk Early-stage Triple-negative Breast Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry); Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE-202012
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Carcinoma Breast; Triple-negative Breast Cancer; Invasive Ductal Carcinoma, Breast
Keywords: Huaier Granule; Triple-negative Breast Cancer; Invasive Ductal Carcinoma, Breast; Adjuvant Treatment
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Carcinoma, Ductal, Breast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huaier Granule + Conventional Treatment/visit (Experimental): Huaier Granule: oral administration, 20g each time, 3 times a day. The starting time of Huaier granule: from the beginning of adjuvant therapy to the end of adjuvant therapy, and within 60 days after the end of adjuvant therapy is also acceptable.
  Conventional Treatment/visit：The postoperative adjuvant therapy and visit of TNBC are based on clinical routine.
  Interventions: Drug: Huaier Granule
- Conventional Treatment/visit (No Intervention): Conventional Treatment/visit：The postoperative adjuvant therapy and visit of TNBC are based on clinical routine.

INTERVENTIONS:
Drug: Huaier Granule — The subjects in the experimental group will be treated with Huaier Granule continuously for 2 years or until the disease progressed, intolerable toxicity, withdrawal of informed consent form or died for any reason.
  Other Names: Z20000109（NMPA Approval Number）
  Arms: Huaier Granule + Conventional Treatment/visit

SUMMARY:
This is a prospective, multicenter, randomized, parallel controlled, open-label study. The primary purpose of this study is to evaluate the efficacy of Huaier Granule on postoperative adjuvant therapy of high-risk early-stage triple-negative invasive ductal carcinoma. The Secondary purposes are to evaluate the safety of long-term use of Huaier granules as postoperative adjuvant treatment of high-risk early-stage triple-negative invasive ductal carcinoma, and the changes of quality of life score after treatment with Huaier granule.

DETAILED DESCRIPTION:
Triple-negative breast cancer（TNBC） accounts for 10% to 20% of breast cancer. TNBC is more likely to show lymph node involvement at diagnosis, and biologically more aggressive. Women with TNBC have a higher rate of distant recurrence at early-stage and a worse 5-year prognosis than women of other molecular types. Although PARP inhibitors and immune checkpoint inhibitors are showing promise to patients with advanced TNBC, however, these targeted therapies and immunotherapy for TNBC can not increase the clinical benefits of early-stage patients.

As adjuvant therapy for hepatocellular carcinoma after curative liver resection, a multicentre study demonstrated a significant prolongation of RFS and reduced extrahepatic recurrence in Huaier group. Retrospective studies have shown that Huaier granules can improve the rates of disease-free survival（DFS） and overall survival（OS）, and reduce the incidence of adverse events among operable patients with TNBC.

In this study, 1072 high-risk early-stage triple-negative invasive ductal carcinoma participants (536 cases in the observation group and 536 cases in the control group) from 30 research centers will be included. The block randomization was adopted, participants will be randomly divided into the experimental group (Huaier granule plus conventional treatment/visit) and control group (conventional treatment/visit only). All participants will be followed up for 5 years, including 2-year treatment follow-up and 3-year survival follow-up. During the treatment period, the participants will be followed up every 3 months, and the survival follow-up period will be followed up every 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18 to 70.
2. Histologically confirmed as breast invasive ductal carcinoma.
3. Molecular typing of breast lesions is triple-negative breast cancer, when the patient had multicentric lesions at the same time, all invasive lesions were confirmed as triple-negative.
4. Regional lymph node metastasis confirmed by postoperative pathology [except isolated tumor cells ( ITC )], or tumor response did not achieve pathological complete response (pCR) after neoadjuvant therapy [neoadjuvant chemotherapy completed at least four cycles, the breast has residual invasive cancer or axillary lymph node metastasis ( except isolated tumor cells ) .]
5. There was no local recurrence and distant metastasis of the tumor.
6. The time of randomization is during the postoperative adjuvant therapy or within 60 days after the end of the last postoperative adjuvant therapy.
7. Eastern Cooperative Oncology Group performance status (ECOG PS) ≤ 1.
8. Hepatic function and renal function: serum creatinine level ≤ 1.5 × upper limit of normal (ULN), aspartate aminotransferase (AST) concentration / alanine aminotransferase (ALT) concentration≤ 2.5 × ULN，total serum bilirubin concentration≤ 1.5 × ULN.
9. Blood routine: neutrophil count ≥ 1.5*109 / L, platelet count ≥ 100*109 / L, hemoglobin concentration ≥ 90 g / L (without transfusion).
10. The participants volunteered to join the study with good compliance and signed an informed consent form.

Exclusion Criteria:

1. Bilateral breast cancer.
2. Complicated with severe cardiopathy, hepatopathy, nephropathy, endocrine system diseases. According to the researchers' judgement, the comorbidities can cause unacceptable safety risks and affect participants' compliance with research programs.
3. Suffering from malignant tumors other than breast cancer (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix) in the past 5 years.
4. Allergic to Huaier granule.
5. Pregnant or lactating women, and those who planning a pregnancy during the study period.
6. Participating in other clinical trials or participated in other clinical studies within 3 months.
7. Patients with a poor compliance, or they are not appropriate for this study because of other reasons considered by the researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1072 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-28 (Estimated)

PRIMARY OUTCOMES:
3-year rates of disease-free survival | Start of treatment until 3-year follow-up
  Disease-free survival (DFS)：The time from randomization until the date of the first occurrence of one of the following events: recurrence of ipsilateral invasive breast tumor, local recurrence, distant metastasis, death from any cause, contralateral invasive breast cancer, ipsilateral ductal carcinoma in situ, contralateral ductal carcinoma in situ, second primary invasive carcinoma (except breast cancer).
  3-year rates of disease-free survival: The percentage of participants who have not occurred events described in the DFS definition within 3 years.

SECONDARY OUTCOMES:
3-year rates of overall survival | Start of treatment until 3-year follow-up
  Overall survival (OS): The time from randomization until the date of death from any cause.
  3-year rates of overall survival: The percentage of participants who have not died from any cause within 3 years.
3-year rates of invasive-disease-free survival | Start of treatment until 3-year follow-up
  Invasive-disease-free survival (iDFS): The time from randomization until the date of the first occurrence of one of the following events: recurrence of ipsilateral invasive breast tumor, local recurrence, distant metastasis, death from any cause, contralateral invasive breast cancer, second primary invasive carcinoma (except breast cancer).
  3-year rates of invasive-disease-free survival: The percentage of participants who have not occurred events described in the iDFS definition within 3 years.
5-year rates of disease-free survival | Start of treatment until 5-year follow-up
  5-year rates of disease-free survival: The percentage of participants who have not occurred events described in the DFS definition within 5 years.
5-year rates of overall survival | Start of treatment until 5-year follow-up
  5-year rates of overall survival: The percentage of participants who have not died from any cause within 5 years.
5-year rates of invasive-disease-free survival | Start of treatment until 5-year follow-up
  5-year rates of invasive-disease-free survival: The percentage of participants who have not occurred events described in the iDFS definition within 5 years.
Changes in European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire | Up to 5 years since the start of treatment
  Quality of Life (QOL) will be measured by European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30). The scope of each domain is 0 to 100. Higher scores in the functional and general health areas indicate better functional status and quality of life, and higher scores in the symptomatic areas indicate more symptoms or problems (poorer quality of life).
Incidence and severity of AE or SAE | Start of treatment until 3 year after enrollment
  AE: Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
  SAE: A serious adverse event (experience) or reaction is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Incidence and severity of ADR，SUSAR or SADR | Start of treatment until 3 year after enrollment
  All noxious and unintended responses to a medicinal product related to any dose should be considered adverse drug reactions. A SADR is a serious ADR according to the above criteria of SAE. A SUSAR is an unexpected SADR.

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, PhD, Principal Investigator — Fudan University
Locations (34):
- China (34):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of USTC, Anhui Provincial Hospital, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The Fourth Hospital of Hebei Medical University, Hebei Tumor Hospital, Shijiazhuang, Hebei
  - The First Affiliates Hospital of Ha'erbin University, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Tongji Medical College of HUST, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong Univeristy of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing, Jiangsu
  - Jiangsu Provincial Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - LongHua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'an Jiaotong University (Xibei Hospital), Xi’an, Shanxi
  - The First Affiliatied Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang Univerisity of Medicine, Hangzhou, Zhejiang
  - Huamei Hospital, University of Chinese Academy of Sciences, Ningbo, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - The First School of Medicine, School of Information and Engineering,the First Affiliated Hospital of WMU, Wenzhou, Zhejiang
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: No